CLINICAL TRIAL: NCT02351856
Title: An Open-label Rollover Study of ARRY-371797 in Patients With Symptomatic Genetic Dilated Cardiomyopathy Due to a Lamin A/C Gene Mutation
Brief Title: A Rollover Study of ARRY-371797 in Patients With LMNA-Related Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-797-001; C4411001 (Other: Alias Study Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: LMNA-Related Dilated Cardiomyopathy
Keywords: laminopathy; ARRY-797
MeSH Terms: conditions — Cardiomyopathy, Dilated; Laminopathies | interventions — ARRY-371797

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARRY-371797 (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor, oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor, oral — multiple dose, single schedule

SUMMARY:
This is a rollover study designed to investigate the safety and effectiveness of investigational study drug ARRY-371797 in patients who previously received ARRY-371797 in a study for patients with LMNA-related dilated cardiomyopathy sponsored by Array BioPharma and may, in the Investigator's opinion, derive benefit from continued treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Received ARRY-371797 as treatment for a genetic dilated cardiomyopathy secondary to LMNA mutations in a clinical study sponsored by Array BioPharma.
* May, in the opinion of the Investigator, benefit from continued ARRY-371797 treatment.
* Additional criteria exist.

Key Exclusion Criteria:

* Discontinued treatment in the parent study for any reason other than study completion or Sponsor termination of the study.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - University of Colorado Hospital, Aurora, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Meriter Wisconsin Heart, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Garcia-Pavia P, Palomares JFR, Sinagra G, Barriales-Villa R, Lakdawala NK, Gottlieb RL, Goldberg RI, Elliott P, Lee P, Li H, Angeli FS, Judge DP, MacRae CA; REALM-DCM Investigators. REALM-DCM: A Phase 3, Multinational, Randomized, Placebo-Controlled Trial of ARRY-371797 in Patients With Symptomatic LMNA-Related Dilated Cardiomyopathy. Circ Heart Fail. 2024 Jul;17(7):e011548. doi: 10.1161/CIRCHEARTFAILURE.123.011548. Epub 2024 Jul 9. PMID 38979608
- [Derived] MacRae CA, Taylor MR, Mestroni L, Moses J, Ashley EA, Wheeler MT, Lakdawala NK, Hershberger RE, Sandor V, Saunders ME, Oliver C, Lee PA, Judge DP. Plain Language Summary of Publication of the safety and efficacy of ARRY-371797 in people with dilated cardiomyopathy and a faulty LMNA gene. Future Cardiol. 2023 Feb;19(2):55-63. doi: 10.2217/fca-2022-0099. Epub 2023 Jan 31. PMID 36718638
- [Derived] Judge DP, Lakdawala NK, Taylor MRG, Mestroni L, Li H, Oliver C, Angeli FS, Lee PA, MacRae CA. Long-Term Efficacy and Safety of ARRY-371797 (PF-07265803) in Patients With Lamin A/C-Related Dilated Cardiomyopathy. Am J Cardiol. 2022 Nov 15;183:93-98. doi: 10.1016/j.amjcard.2022.08.001. Epub 2022 Sep 13. PMID 36114020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 8 participants signed the informed consent form (ICF). All were enrolled into the study and assigned to a study treatment. None of them were screen failure.
Groups:
- ARRY-371797: Participants with symptomatic genetic dilated cardiomyopathy due to a LMNA (Gene encoding the Lamin A/C protein) mutation, and who received ARRY-371797 in the parent study, NCT02057341, were enrolled in this rollover study ARRAY-797-001. Participants received ARRY-371797 at the same dose and schedule they were administered at the end of parent study: ARRY-371797 tablet or capsules 400 milligram (mg) twice a day (BID) until treatment discontinuation criteria [withdrawal of consent, unacceptable adverse events (AE) or failure to tolerate ARRY-371797, pregnancy or initiation of breastfeeding, lost to follow-up] were met, (up to a maximum of 282 weeks). If participant had tolerability concerns at 400 mg BID, they were down-titrated to 200 mg BID (400 mg total daily dose). If participant had tolerability concerns at 200 mg BID, they were down-titrated to 100 mg BID (200 mg total daily dose). Participants were followed up to 30 days for safety after last dose of study drug.
Period: Overall Study
Arm/Group | ARRY-371797
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Physician Decision | 5
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- ARRY-371797: Participants with symptomatic genetic dilated cardiomyopathy due to a LMNA mutation, and who received ARRY-371797 in the parent study, NCT02057341, were enrolled in this rollover study ARRAY-797-001. Participants received ARRY-371797 at the same dose and schedule they were administered at the end of parent study: ARRY-371797 tablet or capsules 400 mg BID until treatment discontinuation criteria [withdrawal of consent, unacceptable AE or failure to tolerate ARRY-371797, pregnancy or initiation of breastfeeding, lost to follow-up] were met, (up to a maximum of 282 weeks). If participant had tolerability concerns at 400 mg BID, they were down-titrated to 200 mg BID (400 mg total daily dose). If participant had tolerability concerns at 200 mg BID, they were down-titrated to 100 mg BID (200 mg total daily dose). Participants were followed up to 30 days for safety after last dose of study drug.
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between baseline up to 30 days after last dose of study drug (i.e., maximum up to 282 weeks) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 30 days after last dose of study drug (i.e., maximum up to 282 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants
  SAEs | 6
  TEAEs | 8

2. Primary Outcome: Number of Participants With Change From Baseline Value in Clinical Laboratory Hematology Test Results to Worst Value
Description: In this outcome measure, number of participants with baseline laboratory hematology values as per National Cancer Institute Common Terminology Criteria (NCI-CTC) grade (Grade 0= within normal limits, Grade 1=Mild, Grade 2=Moderate, Grade 3= Severe, Grade 4= Life-threatening) and corresponding changes/shift to the worst CTC grades post baseline were presented. Shift data have been reported for hematology parameters: hemoglobin (g/L), platelets (10^9/L), leukocytes (10^9/L), neutrophils (10^9/L), lymphocytes (10^9/L) and eosinophils (10^9/L). Baseline was defined as last non-missing value before the initial administration of study treatment in parent study and worst post-baseline value defined as worst value between first dose of study drug up to the maximum of 282 weeks. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline, Post-Baseline (anytime from first dose of study drug to maximum duration of up to 282 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug. Here, "Number Analyzed" signifies participants evaluable for specific parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants
  Hemoglobin: grade 0 (baseline grade) to post baseline grade 1 | 3
  Hemoglobin: grade 0 (baseline grade) to post baseline grade 2 | 4
  Hemoglobin: grade 0 (baseline grade) to post baseline grade 3 | 1
  Platelets: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 7
  Platelets: grade 0 (baseline grade) to post baseline grade 0 | 6
  Platelets: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 7
  Platelets: grade 0 (baseline grade) to post baseline grade 1 | 1
  Platelets: grade 1 (baseline grade) to post baseline grade 3: number analyzed (Participants) | 1
  Platelets: grade 1 (baseline grade) to post baseline grade 3 | 1
  Leukocytes: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 6
  Leukocytes: grade 0 (baseline grade) to post baseline grade 0 | 6
  Leukocytes: grade 1 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 2
  Leukocytes: grade 1 (baseline grade) to post baseline grade 1 | 2
  Neutrophils: grade 0 (baseline grade) to post baseline grade 0 | 6
  Neutrophils: grade 0 (baseline grade) to post baseline grade 1 | 2
  Lymphocytes: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 7
  Lymphocytes: grade 0 (baseline grade) to post baseline grade 0 | 6
  Lymphocytes: grade 0 (baseline grade) to post baseline grade 2: number analyzed (Participants) | 7
  Lymphocytes: grade 0 (baseline grade) to post baseline grade 2 | 1
  Lymphocytes: grade 1 (baseline grade) to post baseline grade 2: number analyzed (Participants) | 1
  Lymphocytes: grade 1 (baseline grade) to post baseline grade 2 | 1
  Eosinophils: grade 0 (baseline grade) to post baseline grade 0 | 8

3. Primary Outcome: Number of Participants With Change From Baseline Value in Clinical Laboratory Chemistry Test Results to Worst Value
Description: In this outcome measure, number of participants with baseline laboratory chemistry values as per NCI-CTC grade (Grade 0= within normal limits, Grade 1=Mild, Grade 2=Moderate, Grade 3= Severe, Grade 4= Life-threatening) and corresponding changes/shift to the worst CTC grades post baseline were presented. Shift data have been reported for laboratory parameters: alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, international unit per liter (IU/L), albumin, bilirubin, urea nitrogen, calcium, creatinine, glucose, magnesium, protein and phosphate grams per deciliter (g/dL), potassium and sodium, millimol per liter (mmol/L). Baseline was defined as last non-missing value before the initial administration of study treatment in parent study and worst post-baseline value defined as worst value between first dose of study drug up to the maximum of 282 weeks. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline, Post-Baseline (anytime from first dose of study drug to maximum duration of up to 282 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants
  Alanine aminotransferase: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 7
  Alanine aminotransferase: grade 0 (baseline grade) to post baseline grade 0 | 6
  Alanine aminotransferase: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 7
  Alanine aminotransferase: grade 0 (baseline grade) to post baseline grade 1 | 1
  Alanine aminotransferase: grade 1 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 1
  Alanine aminotransferase: grade 1 (baseline grade) to post baseline grade 1 | 1
  Albumin: grade 0 (baseline grade) to post baseline grade 0 | 7
  Albumin: grade 0 (baseline grade) to post baseline grade 1 | 1
  Alkaline phosphatase: grade 0 (baseline grade) to post baseline grade 0 | 8
  Aspartate aminotransferase: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 5
  Aspartate aminotransferase: grade 0 (baseline grade) to post baseline grade 0 | 3
  Aspartate aminotransferase: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 5
  Aspartate aminotransferase: grade 0 (baseline grade) to post baseline grade 1 | 2
  Aspartate aminotransferase: grade 1 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 3
  Aspartate aminotransferase: grade 1 (baseline grade) to post baseline grade 0 | 3
  Bilirubin: grade 0 (baseline grade) to post baseline grade 0 | 5
  Bilirubin: grade 0 (baseline grade) to post baseline grade 1 | 2
  Bilirubin: grade 0 (baseline grade) to post baseline grade 3 | 1
  Urea nitrogen: grade 0 (baseline grade) to post baseline grade 0 | 4
  Urea nitrogen: grade 0 (baseline grade) to post baseline grade 1 | 3
  Urea nitrogen: grade 0 (baseline grade) to post baseline grade 3 | 1
  Calcium: grade 0 (baseline grade) to post baseline grade 0 | 6
  Calcium: grade 0 (baseline grade) to post baseline grade 1 | 1
  Calcium: grade 0 (baseline grade) to post baseline grade 2 | 1
  Creatinine: grade 0 (baseline grade) to post baseline grade 0 | 7
  Creatinine: grade 0 (baseline grade) to post baseline grade 2 | 1
  Glucose: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 6
  Glucose: grade 0 (baseline grade) to post baseline grade 0 | 3
  Glucose: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 6
  Glucose: grade 0 (baseline grade) to post baseline grade 1 | 2
  Glucose: grade 0 (baseline grade) to post baseline grade 2: number analyzed (Participants) | 6
  Glucose: grade 0 (baseline grade) to post baseline grade 2 | 1
  Glucose: grade 1 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 1
  Glucose: grade 1 (baseline grade) to post baseline grade 0 | 1
  Glucose: grade 2 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 1
  Glucose: grade 2 (baseline grade) to post baseline grade 1 | 1
  Magnesium: grade 0 (baseline grade) to post baseline grade 0 | 8
  Phosphate: grade 0 (baseline grade) to post baseline grade 0 | 5
  Phosphate: grade 0 (baseline grade) to post baseline grade 1 | 2
  Phosphate: grade 0 (baseline grade) to post baseline grade 3 | 1
  Potassium: grade 0 (baseline grade) to post baseline grade 0 | 6
  Potassium: grade 0 (baseline grade) to post baseline grade 1 | 2
  Protein: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 7
  Protein: grade 0 (baseline grade) to post baseline grade 0 | 3
  Protein: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 7
  Protein: grade 0 (baseline grade) to post baseline grade 1 | 3
  Protein: grade 0 (baseline grade) to post baseline grade 3: number analyzed (Participants) | 7
  Protein: grade 0 (baseline grade) to post baseline grade 3 | 1
  Protein: grade 1 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 1
  Protein: grade 1 (baseline grade) to post baseline grade 1 | 1
  Sodium: grade 0 (baseline grade) to post baseline grade 0: number analyzed (Participants) | 7
  Sodium: grade 0 (baseline grade) to post baseline grade 0 | 5
  Sodium: grade 0 (baseline grade) to post baseline grade 1: number analyzed (Participants) | 7
  Sodium: grade 0 (baseline grade) to post baseline grade 1 | 2
  Sodium: grade 2 (baseline grade) to post baseline grade 2 | 1

4. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included the assessment of skin, head, ears, eyes, nose, throat, cardiovascular system, abdomen and lungs. Abnormality in physical examination were based on investigator's discretion.
Time Frame: Baseline up to 30 days after last dose of study drug (i.e., maximum up to 282 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants | 8

5. Primary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Following vital signs parameters were analyzed using prespecified range of results for signs of clinical significance: systolic blood pressure in millimeters of mercury (mmHg): <90 mmHg and ≥160 mmHg, diastolic blood pressure: <60 mmHg and ≥100 mmHg, heart rate in beats per minute (bpm): <40bpm and >120 bpm, temperature in degree Celsius (C): <36.1 and > 37.2 degree C.
Time Frame: Baseline up to 30 days after last dose of study drug (i.e., maximum up to 282 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants | 6

6. Primary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: Following ECG parameters were analyzed using prespecified range of results for signs of clinical significance: heart rate: <40bpm and >120 bpm; QT/QTcF (QT interval corrected using Fridericia's formula) criteria: QT interval >500 ms; QTcF interval >450 ms; or change from baseline in QTcF >30 ms.
Time Frame: Baseline up to 30 days after last dose of study drug (i.e., maximum up to 282 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Participants | 8

7. Secondary Outcome: Change From Baseline in Six Minute Walk Test (6MWT) Distance at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: 6MWT was the distance that a participant could quickly walk on a flat, hard surface in a period of 6 minutes. Participants were asked to walk a set course of 30 meters for 6 minutes (timed), and the distance walked (in meters) was recorded. Change from baseline in 6MWT distance at specified time points were reported. Baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: Baseline, Day 1, Weeks 24, 48, 72, 96 and early termination visit (anytime within the maximum duration of up to 282 weeks)
Population: Efficacy analysis set included participants who had at least 1 post-baseline efficacy evaluation. Here, "Number Analyzed" signifies participants evaluable for specific time point.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Meters
  Baseline | 319.5 (48.48)
  Change at Day 1 | 55.3 (51.92)
  Change at Week 24: number analyzed (Participants) | 6
  Change at Week 24 | 32.2 (62.31)
  Change at Week 48: number analyzed (Participants) | 4
  Change at Week 48 | 55.8 (63.76)
  Change at Week 72: number analyzed (Participants) | 5
  Change at Week 72 | 42.6 (74.92)
  Change at Week 96: number analyzed (Participants) | 5
  Change at Week 96 | 10.8 (113.12)
  Change at Early Termination Visit: number analyzed (Participants) | 4
  Change at Early Termination Visit | -14.3 (68.78)

8. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Index (LVESVI) and Left Ventricular End Diastolic Volume Index (LVEDVI) at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: LVESVI and LVEDVI were echocardiographic assessment of left ventricular remodeling. Baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milliliter per meter square
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Milliliter per meter square
  LVESVI: Baseline | 45.25 (12.766)
  LVESVI: change at Day 1: number analyzed (Participants) | 6
  LVESVI: change at Day 1 | 1.83 (7.932)
  LVESVI: change at Week 24: number analyzed (Participants) | 5
  LVESVI: change at Week 24 | -0.01 (5.403)
  LVESVI: change at Week 48: number analyzed (Participants) | 4
  LVESVI: change at Week 48 | -1.31 (11.707)
  LVESVI: change at Week 72: number analyzed (Participants) | 5
  LVESVI: change at Week 72 | -1.36 (14.374)
  LVESVI: change at Week 96: number analyzed (Participants) | 5
  LVESVI: change at Week 96 | -0.39 (4.090)
  LVESVI: change at Early Termination Visit: number analyzed (Participants) | 3
  LVESVI: change at Early Termination Visit | -0.26 (4.447)
  LVEDVI: Baseline | 70.41 (13.933)
  LVEDVI: change at Day 1: number analyzed (Participants) | 6
  LVEDVI: change at Day 1 | 2.31 (11.504)
  LVEDVI: change at Week 24: number analyzed (Participants) | 5
  LVEDVI: change at Week 24 | 1.19 (12.320)
  LVEDVI: change at Week 48: number analyzed (Participants) | 4
  LVEDVI: change at Week 48 | -1.13 (9.338)
  LVEDVI: change at Week 72: number analyzed (Participants) | 5
  LVEDVI: change at Week 72 | -2.99 (14.063)
  LVEDVI: change at Week 96: number analyzed (Participants) | 5
  LVEDVI: change at Week 96 | -1.54 (13.236)
  LVEDVI: change at Early Termination Visit: number analyzed (Participants) | 3
  LVEDVI: change at Early Termination Visit | 6.36 (7.089)

9. Secondary Outcome: Change From Baseline in Left Ventricular Mass (LVM) at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: LVM is the weight of the left ventricle in grams estimated by echocardiography. For this outcome measure, Baseline is the pre-dose baseline of parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Grams
  Baseline: number analyzed (Participants) | 7
  Baseline | 169.97 (65.592)
  Change at Day 1: number analyzed (Participants) | 7
  Change at Day 1 | 4.38 (39.217)
  Change at Week 24: number analyzed (Participants) | 6
  Change at Week 24 | 12.39 (31.789)
  Change at Week 48: number analyzed (Participants) | 5
  Change at Week 48 | 7.46 (32.190)
  Change at Week 72: number analyzed (Participants) | 5
  Change at Week 72 | 20.87 (43.152)
  Change at Week 96: number analyzed (Participants) | 5
  Change at Week 96 | 15.25 (33.332)
  Change at Early Termination Visit: number analyzed (Participants) | 3
  Change at Early Termination Visit | 8.97 (14.194)

10. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: LVEF was the fraction of the end-diastolic volume (EDV) that was ejected out of left ventricle with each contraction, estimated by echocardiography. EDV was the volume of blood within a ventricle immediately before a contraction. Baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of EDV
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Percentage of EDV
  Baseline | 37.88 (10.633)
  Change at Day 1: number analyzed (Participants) | 7
  Change at Day 1 | 0.10 (5.322)
  Change at Week 24: number analyzed (Participants) | 6
  Change at Week 24 | 1.50 (5.032)
  Change at Week 48: number analyzed (Participants) | 5
  Change at Week 48 | 0.10 (7.195)
  Change at Week 72: number analyzed (Participants) | 5
  Change at Week 72 | 4.27 (7.882)
  Change at Week 96: number analyzed (Participants) | 4
  Change at Week 96 | 1.71 (3.538)
  Change at Early Termination Visit: number analyzed (Participants) | 3
  Change at Early Termination Visit | 2.11 (4.137)

11. Secondary Outcome: Change From Baseline in Left Ventricular Mass (LVM) to Volume Ratio at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: LVM divided by the end diastolic volume, estimated by echocardiography. Baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Grams per milliliter
  Baseline: number analyzed (Participants) | 7
  Baseline | 1.32 (0.568)
  Change at Day 1: number analyzed (Participants) | 6
  Change at Day 1 | -0.04 (0.357)
  Change at Week 24: number analyzed (Participants) | 5
  Change at Week 24 | 0.03 (0.259)
  Change at Week 48: number analyzed (Participants) | 4
  Change at Week 48 | 0.05 (0.137)
  Change at Week 72: number analyzed (Participants) | 4
  Change at Week 72 | 0.14 (0.295)
  Change at Week 96: number analyzed (Participants) | 4
  Change at Week 96 | 0.21 (0.442)
  Change at Early Termination Visit: number analyzed (Participants) | 3
  Change at Early Termination Visit | 0.08 (0.378)

12. Secondary Outcome: Change From Baseline in Right Ventricular End Diastolic Diameter at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: The internal diameter of the right ventricle at the end of diastole, measured by echocardiography. Baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Centimeter
  Baseline | 3.79 (0.686)
  Change at Day 1: number analyzed (Participants) | 6
  Change at Day 1 | 0.30 (0.329)
  Change at Week 24: number analyzed (Participants) | 6
  Change at Week 24 | 0.02 (0.635)
  Change at Week 48 | 0.59 (0.462)
  Change at Week 72 | 0.14 (0.604)
  Change at Week 96: number analyzed (Participants) | 5
  Change at Week 96 | 0.26 (0.853)
  Change at Early Termination Visit: number analyzed (Participants) | 2
  Change at Early Termination Visit | 1.15 (1.909)

13. Secondary Outcome: Change From Baseline in Right Ventricular Fractional Area at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: Right ventricular fractional area change is a measure of global right ventricular systolic function estimated by echocardiography. For this outcome measure, Baseline is the pre-dose baseline of parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Percentage
  Baseline | 22.14 (6.896)
  Change at Day 1: number analyzed (Participants) | 6
  Change at Day 1 | 8.25 (10.252)
  Change at Week 24: number analyzed (Participants) | 6
  Change at Week 24 | 8.67 (13.358)
  Change at Week 48: number analyzed (Participants) | 5
  Change at Week 48 | 7.85 (13.051)
  Change at Week 72: number analyzed (Participants) | 5
  Change at Week 72 | 8.22 (12.059)
  Change at Week 96: number analyzed (Participants) | 5
  Change at Week 96 | 1.95 (6.945)
  Change at Early Termination Visit: number analyzed (Participants) | 2
  Change at Early Termination Visit | 0.51 (8.004)

14. Secondary Outcome: Change From Baseline in 36-Item Short-Form (SF-36) Health Survey Score at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: The SF-36 health survey is a participant-reported survey to measure participant's health. It is a 36-item questionnaire used to measure 8 various aspects of health (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health). The score range for each of the 8 aspects was from 0 (maximum disability) to 100 (no disability), higher scores indicating good health condition. For this analysis, baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Units on a scale
  Vitality: Baseline | 39.97 (11.858)
  Vitality: change at Day 1 | -0.74 (7.901)
  Vitality: change at Week 24: number analyzed (Participants) | 6
  Vitality: change at Week 24 | -0.50 (8.491)
  Vitality: change at Week 48: number analyzed (Participants) | 4
  Vitality: change at Week 48 | -2.97 (8.405)
  Vitality: change at Week 72: number analyzed (Participants) | 5
  Vitality: change at Week 72 | -3.57 (8.246)
  Vitality: change at Week 96 | -5.94 (8.403)
  Vitality: change at Early Termination Visit: number analyzed (Participants) | 5
  Vitality: change at Early Termination Visit | -1.78 (7.462)
  Physical functioning: Baseline | 35.77 (9.540)
  Physical functioning: change at Day 1 | -0.24 (6.508)
  Physical functioning: change at Week 24: number analyzed (Participants) | 6
  Physical functioning: change at Week 24 | 0.96 (6.929)
  Physical functioning: change at Week 48: number analyzed (Participants) | 5
  Physical functioning: change at Week 48 | -1.15 (10.539)
  Physical functioning: change at Week 72: number analyzed (Participants) | 5
  Physical functioning: change at Week 72 | 0.77 (5.347)
  Physical functioning: change at Week 96: number analyzed (Participants) | 5
  Physical functioning: change at Week 96 | 1.53 (7.944)
  Physical functioning: change at Early Termination Visit: number analyzed (Participants) | 5
  Physical functioning: change at Early Termination Visit | -6.51 (5.512)
  Bodily pain: Baseline | 51.11 (8.635)
  Bodily pain: change at Day 1 | -1.92 (9.561)
  Bodily pain: change at Week 24: number analyzed (Participants) | 6
  Bodily pain: change at Week 24 | -3.97 (10.195)
  Bodily pain: change at Week 48: number analyzed (Participants) | 4
  Bodily pain: change at Week 48 | 2.72 (8.076)
  Bodily pain: change at Week 72: number analyzed (Participants) | 5
  Bodily pain: change at Week 72 | 3.06 (4.648)
  Bodily pain: change at Week 96: number analyzed (Participants) | 5
  Bodily pain: change at Week 96 | -4.27 (5.991)
  Bodily pain: change at Early Termination Visit: number analyzed (Participants) | 5
  Bodily pain: change at Early Termination Visit | -5.56 (10.725)
  General health: Baseline | 36.37 (8.372)
  General health: change at Day 1 | 1.78 (5.637)
  General health: change at Week 24: number analyzed (Participants) | 6
  General health: change at Week 24 | 0 (3.669)
  General health: change at Week 48: number analyzed (Participants) | 5
  General health: change at Week 48 | -2.09 (8.717)
  General health: change at Week 72: number analyzed (Participants) | 5
  General health: change at Week 72 | -1.43 (8.057)
  General health: change at Week 96: number analyzed (Participants) | 5
  General health: change at Week 96 | -1.62 (8.612)
  General health: change at Early Termination Visit: number analyzed (Participants) | 5
  General health: change at Early Termination Visit | 1.90 (4.801)
  Role physical: Baseline | 32.74 (8.691)
  Role physical: change at Day 1 | 5.61 (8.315)
  Role physical: change at Week 24: number analyzed (Participants) | 6
  Role physical: change at Week 24 | 4.49 (9.420)
  Role physical: change at Week 48: number analyzed (Participants) | 4
  Role physical: change at Week 48 | 5.62 (6.982)
  Role physical: change at Week 72: number analyzed (Participants) | 5
  Role physical: change at Week 72 | 9.43 (4.316)
  Role physical: change at Week 96: number analyzed (Participants) | 5
  Role physical: change at Week 96 | 2.25 (8.249)
  Role physical: change at Early Termination Visit: number analyzed (Participants) | 5
  Role physical: change at Early Termination Visit | 4.94 (12.339)
  Role emotional: Baseline | 43.98 (11.772)
  Role emotional: change at Day 1 | 1.74 (8.325)
  Role emotional: change at Week 24: number analyzed (Participants) | 6
  Role emotional: change at Week 24 | 0.00 (7.940)
  Role emotional: change at Week 48: number analyzed (Participants) | 4
  Role emotional: change at Week 48 | -3.48 (14.773)
  Role emotional: change at Week 72: number analyzed (Participants) | 5
  Role emotional: change at Week 72 | 5.57 (12.696)
  Role emotional: change at Week 96: number analyzed (Participants) | 5
  Role emotional: change at Week 96 | -6.96 (18.095)
  Role emotional: change at Early Termination Visit: number analyzed (Participants) | 5
  Role emotional: change at Early Termination Visit | 0.00 (8.532)
  Social functioning: Baseline | 41.05 (9.936)
  Social functioning: change at Day 1 | -1.26 (12.778)
  Social functioning: change at Week 24: number analyzed (Participants) | 6
  Social functioning: change at Week 24 | 1.67 (11.285)
  Social functioning: change at Week 48: number analyzed (Participants) | 4
  Social functioning: change at Week 48 | -2.51 (8.683)
  Social functioning: change at Week 72: number analyzed (Participants) | 5
  Social functioning: change at Week 72 | 3.01 (7.605)
  Social functioning: change at Week 96: number analyzed (Participants) | 5
  Social functioning: change at Week 96 | -3.01 (9.106)
  Social functioning: change at Early Termination Visit: number analyzed (Participants) | 5
  Social functioning: change at Early Termination Visit | -4.01 (9.641)
  Mental health: Baseline | 47.60 (14.378)
  Mental health: change at Day 1 | 2.94 (3.816)
  Mental health: change at Week 24: number analyzed (Participants) | 6
  Mental health: change at Week 24 | -0.43 (7.654)
  Mental health: change at Week 48: number analyzed (Participants) | 4
  Mental health: change at Week 48 | -5.23 (7.702)
  Mental health: change at Week 72: number analyzed (Participants) | 5
  Mental health: change at Week 72 | -2.09 (15.405)
  Mental health: change at Week 96: number analyzed (Participants) | 5
  Mental health: change at Week 96 | -4.71 (14.373)
  Mental health: change at Early Termination Visit: number analyzed (Participants) | 5
  Mental health: change at Early Termination Visit | 0 (7.623)
  Mental Classification System (MCS): Baseline | 46.96 (13.995)
  MCS: change at Day 1 | 1.19 (6.558)
  MCS: change at Week 24: number analyzed (Participants) | 6
  MCS: change at Week 24 | -0.27 (8.294)
  MCS: change at Week 48: number analyzed (Participants) | 4
  MCS: change at Week 48 | -7.07 (10.751)
  MCS: change at Week 72: number analyzed (Participants) | 5
  MCS: change at Week 72 | -0.24 (15.610)
  MCS: change at Week 96: number analyzed (Participants) | 5
  MCS: change at Week 96 | -7.70 (14.765)
  MCS: change at Early Termination Visit: number analyzed (Participants) | 5
  MCS: change at Early Termination Visit | -0.10 (7.394)
  Physical Classification System (PCS): Baseline | 36.32 (8.201)
  PCS: change at Day 1 | 0.71 (7.519)
  PCS: change at Week 24: number analyzed (Participants) | 6
  PCS: change at Week 24 | 0.79 (7.552)
  PCS: change at Week 48: number analyzed (Participants) | 4
  PCS: change at Week 48 | 6.19 (1.535)
  PCS: change at Week 72: number analyzed (Participants) | 5
  PCS: change at Week 72 | 3.52 (5.672)
  PCS: change at Week 96: number analyzed (Participants) | 5
  PCS: change at Week 96 | 1.90 (5.656)
  PCS: change at Early Termination Visit: number analyzed (Participants) | 5
  PCS: change at Early Termination Visit | -2.34 (6.730)

15. Secondary Outcome: Change From Baseline in Quality of Life by Kansas City Cardiomyopathy Questionnaire (KCCQ) Scores at Day 1, Weeks 24, 48, 72, 96 and Early Termination Visit
Description: KCCQ was a 23-item heart failure specific questionnaire quantified into following 10 summary scores: physical limitation score, symptom frequency score, symptom severity score, symptom stability score, total symptoms score, quality of life score, social interference score, self-efficacy score, overall summary score and clinical summary score. These scores ranged from 0 to 100, where higher scores indicated better functioning, fewer symptoms, and better disease specific quality of life. For this analysis, baseline was defined as last non-missing value before the initial administration of study treatment in parent study.
Time Frame: as for outcome 7
Population: Efficacy analysis set was included participants who had at least 1 post-Baseline efficacy evaluation. Here, "Number Analyzed" signifies participants evaluable for specific time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ARRY-371797
Number analyzed (Participants) | 8
Units on a scale
  Physical limitation score: Baseline | 60.42 (27.186)
  Physical limitation score: change at Day 1: number analyzed (Participants) | 7
  Physical limitation score: change at Day 1 | 0.60 (15.296)
  Physical limitation score: change at Week 24: number analyzed (Participants) | 6
  Physical limitation score: change at Week 24 | 8.33 (19.365)
  Physical limitation score: change at Week 48: number analyzed (Participants) | 5
  Physical limitation score: change at Week 48 | -0.83 (27.386)
  Physical limitation score: change at Week 72: number analyzed (Participants) | 5
  Physical limitation score: change at Week 72 | 13.83 (23.204)
  Physical limitation score: change at Week 96: number analyzed (Participants) | 5
  Physical limitation score: change at Week 96 | 12.17 (23.545)
  Physical limitation score: change at Early Termination Visit: number analyzed (Participants) | 4
  Physical limitation score: change at Early Termination Visit | -8.33 (6.804)
  Symptom stability score: Baseline | 53.13 (8.839)
  Symptom stability score: change at Day 1 | 0 (13.363)
  Symptom stability score: change at Week 24: number analyzed (Participants) | 6
  Symptom stability score: change at Week 24 | 4.17 (24.580)
  Symptom stability score: change at Week 48: number analyzed (Participants) | 5
  Symptom stability score: change at Week 48 | -5.00 (11.180)
  Symptom stability score: change at Week 72: number analyzed (Participants) | 5
  Symptom stability score: change at Week 72 | 5.00 (27.386)
  Symptom stability score: change at Week 96: number analyzed (Participants) | 5
  Symptom stability score: change at Week 96 | -15.00 (13.693)
  Symptom stability score: change at Early Termination Visit: number analyzed (Participants) | 5
  Symptom stability score: change at Early Termination Visit | -5.00 (11.180)
  Symptom frequency score: Baseline | 73.18 (20.334)
  Symptom frequency score: change at Day 1 | -1.30 (10.018)
  Symptom frequency score: change at Week 24: number analyzed (Participants) | 6
  Symptom frequency score: change at Week 24 | -4.86 (18.942)
  Symptom frequency score: change at Week 48: number analyzed (Participants) | 5
  Symptom frequency score: change at Week 48 | -19.17 (27.418)
  Symptom frequency score: change at Week 72: number analyzed (Participants) | 5
  Symptom frequency score: change at Week 72 | -3.33 (13.060)
  Symptom frequency score: change at Week 96: number analyzed (Participants) | 5
  Symptom frequency score: change at Week 96 | -17.50 (21.123)
  Symptom frequency score: change at Early Termination Visit: number analyzed (Participants) | 5
  Symptom frequency score: change at Early Termination Visit | -7.92 (9.592)
  Symptom burden score: Baseline | 72.92 (21.708)
  Symptom burden score: change at Day 1 | -1.04 (10.387)
  Symptom burden score: change at Week 24: number analyzed (Participants) | 6
  Symptom burden score: change at Week 24 | -2.78 (11.386)
  Symptom burden score: change at Week 48: number analyzed (Participants) | 5
  Symptom burden score: change at Week 48 | -16.67 (17.678)
  Symptom burden score: change at Week 72: number analyzed (Participants) | 5
  Symptom burden score: change at Week 72 | 5.00 (20.069)
  Symptom burden score: change at Week 96: number analyzed (Participants) | 5
  Symptom burden score: change at Week 96 | -15.00 (29.107)
  Symptom burden score: change at Early Termination Visit: number analyzed (Participants) | 5
  Symptom burden score: change at Early Termination Visit | -6.67 (14.907)
  Total symptom score: Baseline | 73.05 (20.672)
  Total symptom score: change at Day 1 | -1.17 (9.858)
  Total symptom score: change at Week 24: number analyzed (Participants) | 6
  Total symptom score: change at Week 24 | -3.82 (15.004)
  Total symptom score: change at Week 48: number analyzed (Participants) | 5
  Total symptom score: change at Week 48 | -17.92 (22.467)
  Total symptom score: change at Week 72: number analyzed (Participants) | 5
  Total symptom score: change at Week 72 | 0.83 (15.084)
  Total symptom score: change at Week 96: number analyzed (Participants) | 5
  Total symptom score: change at Week 96 | -16.25 (24.358)
  Total symptom score: change at Early Termination Visit: number analyzed (Participants) | 5
  Total symptom score: change at Early Termination Visit | -7.29 (10.725)
  Self-efficacy score: Baseline | 85.94 (12.388)
  Self-efficacy score: change at Day 1 | 6.25 (11.573)
  Self-efficacy score: change at Week 24: number analyzed (Participants) | 6
  Self-efficacy score: change at Week 24 | 2.08 (16.615)
  Self-efficacy score: change at Week 48: number analyzed (Participants) | 5
  Self-efficacy score: change at Week 48 | 5.00 (11.180)
  Self-efficacy score: change at Week 72: number analyzed (Participants) | 5
  Self-efficacy score: change at Week 72 | 7.50 (14.252)
  Self-efficacy score: change at Week 96: number analyzed (Participants) | 5
  Self-efficacy score: change at Week 96 | 10.00 (10.458)
  Self-efficacy score: change at Early Termination Visit: number analyzed (Participants) | 5
  Self-efficacy score: change at Early Termination Visit | 7.50 (11.180)
  Quality of life score: Baseline | 52.08 (28.781)
  Quality of life score: change at Day 1 | 7.29 (16.925)
  Quality of life score: change at Week 24: number analyzed (Participants) | 6
  Quality of life score: change at Week 24 | 4.17 (13.693)
  Quality of life score: change at Week 48: number analyzed (Participants) | 5
  Quality of life score: change at Week 48 | -13.33 (21.731)
  Quality of life score: change at Week 72: number analyzed (Participants) | 5
  Quality of life score: change at Week 72 | 10.00 (25.954)
  Quality of life score: change at Week 96: number analyzed (Participants) | 5
  Quality of life score: change at Week 96 | -5.00 (28.626)
  Quality of life score: change at Early Termination Visit | 13.33 (33.124)
  Social limitation score: Baseline | 57.81 (29.267)
  Social limitation score: change at Day 1 | 10.16 (21.635)
  Social limitation score: change at Week 24: number analyzed (Participants) | 6
  Social limitation score: change at Week 24 | 3.47 (26.506)
  Social limitation score: change at Week 48: number analyzed (Participants) | 4
  Social limitation score: change at Week 48 | -9.38 (10.825)
  Social limitation score: change at Week 72: number analyzed (Participants) | 5
  Social limitation score: change at Week 72 | 9.17 (18.669)
  Social limitation score: change at Week 96: number analyzed (Participants) | 4
  Social limitation score: change at Week 96 | -11.46 (18.980)
  Social limitation score: change at Early Termination Visit: number analyzed (Participants) | 4
  Social limitation score: change at Early Termination Visit | 1.56 (29.920)
  Overall summary score: Baseline | 60.84 (25.603)
  Overall summary score: change at Day 1 | 4.74 (13.906)
  Overall summary score: change at Week 24: number analyzed (Participants) | 6
  Overall summary score: change at Week 24 | 3.04 (14.082)
  Overall summary score: change at Week 48: number analyzed (Participants) | 5
  Overall summary score: change at Week 48 | -12.64 (21.030)
  Overall summary score: change at Week 72: number analyzed (Participants) | 5
  Overall summary score: change at Week 72 | 8.46 (19.155)
  Overall summary score: change at Week 96: number analyzed (Participants) | 5
  Overall summary score: change at Week 96 | -3.76 (22.697)
  Overall summary score: change at Early Termination Visit: number analyzed (Participants) | 5
  Overall summary score: change at Early Termination Visit | 2.55 (19.283)
  Clinical summary score: Baseline | 66.73 (23.833)
  Clinical summary score: change at Day 1 | 0.33 (11.729)
  Clinical summary score: change at Week 24: number analyzed (Participants) | 6
  Clinical summary score: change at Week 24 | 2.26 (13.955)
  Clinical summary score: change at Week 48: number analyzed (Participants) | 5
  Clinical summary score: change at Week 48 | -9.38 (22.619)
  Clinical summary score: change at Week 72: number analyzed (Participants) | 5
  Clinical summary score: change at Week 72 | 7.33 (18.803)
  Clinical summary score: change at Week 96: number analyzed (Participants) | 5
  Clinical summary score: change at Week 96 | -2.04 (22.629)
  Clinical summary score: change at Early Termination Visit: number analyzed (Participants) | 5
  Clinical summary score: change at Early Termination Visit | -5.10 (9.521)

16. Secondary Outcome: Mean Plasma Concentration of ARRY-371797 and Metabolites (AR00420643, AR00428028, AR00486705)
Description: Plasma concentrations of ARRY-371797 and its metabolites (AR00420643, AR00428028 and AR00486705) was summarized on Day 1, Weeks 12 and 24 at both pre and post dose.
Time Frame: Pre dose and post dose on Day 1, Weeks 12 and 24
Population: Pharmacokinetic (PK) analysis set included all participants who had at least 1 plasma sample with associated PK concentration results. Here, "Number Analyzed" signifies participants evaluable at specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | ARRY-371797
Number analyzed (Participants) | 7
Nanogram per milliliter
  ARRY-371797 Day 1 (Pre-dose): number analyzed (Participants) | 6
  ARRY-371797 Day 1 (Pre-dose) | 4.7136 (209.88)
  ARRY-371797 Day 1 (Post-dose) | 54.053 (643.32)
  ARRY-371797 Week 12 (Pre-dose): number analyzed (Participants) | 3
  ARRY-371797 Week 12 (Pre-dose) | 3.9258 (155.51)
  ARRY-371797 Week 12 (Post-dose): number analyzed (Participants) | 6
  ARRY-371797 Week 12 (Post-dose) | 109.10 (205.28)
  ARRY-371797 Week 24 (Pre-dose): number analyzed (Participants) | 4
  ARRY-371797 Week 24 (Pre-dose) | 4.9345 (300.53)
  ARRY-371797 Week 24 (Post-dose): number analyzed (Participants) | 5
  ARRY-371797 Week 24 (Post-dose) | 41.653 (691.82)
  AR00420643 Day 1 (Pre-dose) | 80.859 (171.38)
  AR00420643 Day 1 (Post-dose) | 348.45 (281.51)
  AR00420643 Week 12 (Pre-dose): number analyzed (Participants) | 5
  AR00420643 Week 12 (Pre-dose) | 33.749 (NA) — Per the decision rules written in the Statistical Analysis Plan (SAP), the number of below the limit of quantitation (BLQ) values for the -643 analyte resulted in geometric coefficient of variation (CV), being not reportable.
  AR00420643 Week 12 (Post-dose): number analyzed (Participants) | 6
  AR00420643 Week 12 (Post-dose) | 432.99 (189.13)
  AR00420643 Week 24 (Pre-dose): number analyzed (Participants) | 5
  AR00420643 Week 24 (Pre-dose) | 73.737 (219.07)
  AR00420643 Week 24 (Post-dose): number analyzed (Participants) | 5
  AR00420643 Week 24 (Post-dose) | 258.80 (411.34)
  AR00428028 Day 1 (Pre-dose) | 44.453 (134.15)
  AR00428028 Day 1 (Post-dose) | 47.392 (110.81)
  AR00428028 Week 12 (Pre-dose): number analyzed (Participants) | 6
  AR00428028 Week 12 (Pre-dose) | 24.003 (131.07)
  AR00428028 Week 12 (Post-dose): number analyzed (Participants) | 6
  AR00428028 Week 12 (Post-dose) | 27.213 (96.919)
  AR00428028 Week 24 (Pre-dose): number analyzed (Participants) | 5
  AR00428028 Week 24 (Pre-dose) | 32.625 (69.620)
  AR00428028 Week 24 (Post-dose): number analyzed (Participants) | 5
  AR00428028 Week 24 (Post-dose) | 32.102 (80.353)
  AR00486705 Day 1 (Pre-dose) | 6.1025 (256.23)
  AR00486705 Day 1 (Post-dose) | 14.541 (256.54)
  AR00486705 Week 12 (Pre-dose): number analyzed (Participants) | 5
  AR00486705 Week 12 (Pre-dose) | 4.0176 (NA) — Per the decision rules written in the SAP, the number of BLQ values for the -643 analyte resulted in geometric CV being not reportable.
  AR00486705 Week 12 (Post-dose): number analyzed (Participants) | 6
  AR00486705 Week 12 (Post-dose) | 13.909 (237.85)
  AR00486705 Week 24 (Pre-dose): number analyzed (Participants) | 5
  AR00486705 Week 24 (Pre-dose) | 6.8860 (97.778)
  AR00486705 Week 24 (Post-dose): number analyzed (Participants) | 5
  AR00486705 Week 24 (Post-dose) | 13.389 (177.04)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (maximum up to 282 weeks)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | ARRY-371797
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARRY-371797 (N=8)
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 4
Colitis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Heart transplant (Surgical and medical procedures) | 1
Orthostatic hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARRY-371797 (N=8)
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
External ear cellulitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lyme disease (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 4
Blood creatinine increased (Investigations) | 1
Coronavirus test positive (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02351856/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT02351856/SAP_001.pdf